CLINICAL TRIAL: NCT02048150
Title: Intra-operative Optical Imaging Utilizing Anti-PSMA (Prostate Specific Membrane Antigen) Fluorescent Antibody During Robotic Assisted Laparoscopic Prostatectomy
Brief Title: Intra-operative Optical Imaging With MDX1201-A488 in Patients With Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13405; NCI-2013-02476 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 13405 (Other: City of Hope Medical Center)
Record Dates: First submitted 2014-01-24; First posted 2014-01-29 (Estimated); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Adenocarcinoma of the Prostate; Stage IIB Prostate Cancer; Stage III Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (MDX1201-A488, IOOI, RALP) (Experimental): Patients receive anti-PSMA monoclonal antibody MDX1201-A488 IV over 30 minutes on day 1 and undergo IOOI during RALP on day 3.
  Interventions: Biological: anti-PSMA monoclonal antibody MDX1201-A488; Procedure: robot-assisted laparoscopic surgery; Other: diffuse optical imaging; Other: pharmacological study; Other: Laboratory Biomarker; Other: Questionnaire

INTERVENTIONS:
Biological: anti-PSMA monoclonal antibody MDX1201-A488 — Given IV
  Other Names: MDX1201; MDX1201-A488
Procedure: robot-assisted laparoscopic surgery — Undergo RALP
Other: diffuse optical imaging — Undergo IOOI
  Other Names: diffuse optical spectroscopy; diffuse optical tomography; DOI; near infrared optical tomography
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: Laboratory Biomarker — Correlative studies
Other: Questionnaire — Ancillary studies

SUMMARY:
This pilot clinical trial studies the best dose of anti-prostate specific membrane antigen (PSMA) monoclonal antibody MDX1201-A488 (MDX1201-A488) given before surgery to aid in visualization of the prostate. Attaching a fluorescence, a substance that emits radiation that is visible, to the anti-PMSA antibody and injecting it into the body may help identify the tumor when specialized microscopes are used.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. Determine the preferred imaging dose (if any), based on image quality and correlation with pathological findings, of intravenously administered MDX1201-A488 in a dose-escalating study (doses of 5 and 15 mg) in patients with moderate to high-risk prostate cancer prior to undergoing robotic assisted laparoscopic prostatectomy (RALP), subject to predetermined safety stopping rules.

SECONDARY OBJECTIVES: I. Correlate intra-operative optical imaging (IOOI) findings with pre-operative magnetic resonance imaging (MRI) findings and clinical staging.

OUTLINE: This is a dose-escalation study. Patients receive anti-PSMA monoclonal antibody MDX1201-A488 intravenously (IV) over 30 minutes on day 1 and undergo IOOI during RALP on day 5.

After completion of study treatment, patients are followed up at 4-7 weeks, 3 months, 6 months, 9 months, and 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate; patients with small cell, neuroendocrine, and transitional cell carcinomas are not eligible
* Patients being considered for RALP and pelvic lymphadenectomy with life expectancy greater than 10 years as determined by treating physician
* Patients with moderate to high-risk disease as defined by D' Amico risk stratification and having at least one of the following:

  * Prostate-specific antigen (PSA) level > 10 ng/ml
  * Gleason score >= 7
  * Clinical stage >= T2c
* Any performance status on the Eastern Cooperative Oncology Group (ECOG)
* Men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation
* Bone scan without evidence of skeletal metastases
* Skeletal x-ray film or MRI confirmation of absent skeletal metastases if bone scan findings are equivocal
* 3Tesla (T) multiparametric MRI of the prostate performed at City of Hope (COH) within 6 week time period prior to surgery; MRI without evidence of bladder neck involvement, rectal wall involvement, or pelvic lymphadenopathy with no nodes > 1 cm
* White blood cell (WBC) within normal limits
* Hemoglobin (hgb) > 10 G/dL
* Platelet count (PLT) > 100 K/uL
* Creatinine clearance within normal limits
* Serum glutamic oxaloacetic transaminase (SGOT) < 1.5 x upper limit of normal (ULN)
* Serum glutamate pyruvate transaminase (SGPT) < 1.5 x ULN
* Bilirubin < 1.5 x ULN
* All subjects must have the ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Patients should not have any uncontrolled illness including ongoing or active infection
* Prior treatment of prostate cancer including brachytherapy, radiation therapy, cryosurgery, high-intensity focused ultrasound (HIFU), or vaccine therapy
* Prior pelvic surgery or radiation
* Urinary incontinence requiring condom catheter use or >= 1 pad/day
* Prior anti-incontinence surgery
* Use of neoadjuvant hormonal manipulation
* History of active co-existing non-prostatic malignancies except basal cell skin cancer or squamous cell skin cancer
* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Ages: 36 Years to 74 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-03-05 (Actual); Primary Completion 2018-05-10 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Imaging ability of anti-PMSA monoclonal antibody MDX1201-A488 | Up to 1 year
  The main fluorescence metric will be the minimum fluorescence observed in 10 sampled high power fields from a single representative cancerous section taken per patient. Other metrics will be the mean fluorescence observed in the 10 sampled high power fields, and the median fluorescence observed. The minimum fluorescence is chosen based on the concept that the primary focus is on observing the fluorescence, and areas of peak fluorescence greatly influence the mean, and also have some influence on the median, yet may be of limited relevance.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Zhumkhawala, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States